CLINICAL TRIAL: NCT02483689
Title: The Evaluation of Pre-incisional and Post-closure Local Anesthetic vs. Normal Saline on Postoperative Pain in Pediatric Appendectomies
Brief Title: Evaluation of Local Anesthetic at Incision Site
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valley Anesthesiology Consultants (Other)
Responsible Party: Principal Investigator, Neil Raj Singhal, Doctor, Valley Anesthesiology Consultants
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-047
Record Dates: First submitted 2015-06-22; First posted 2015-06-29 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Post Operative Pain; Appendicitis
Keywords: Post Operative Pain; Appendicitis; Appendectomy; Local Anesthetic; Saline; Pain Management; Surgery; Recovery
MeSH Terms: conditions — Pain, Postoperative; Appendicitis; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): Patient will be given saline with a maximum of 30 cc either pre-incision: local will be to be given intradermally and onto the peritoneum under direct vision; or post-closure local will be injected intradermally after closure
  Interventions: Other: Pre-Incisional Saline; Other: Post-Closure Saline
- Local (Experimental): Patient will be given a total of 0.5 mL/kg of 0.25% Bupivicaine either pre-incision: local will be to be given intradermally and onto the peritoneum under direct vision; or post-closure local will be injected intradermally after closure
  Interventions: Drug: Pre Incisional Local Anesthetic; Drug: Post-Closure Local Anesthetic

INTERVENTIONS:
Drug: Pre Incisional Local Anesthetic — Patient will be given a total of 0.5 mL/kg of 0.25% Bupivicaine either pre-incision: local will be to be given intradermally and onto the peritoneum under direct vision; or post-closure local will be injected intradermally after closure
  Other Names: Bupivicaine
  Arms: Local
Other: Pre-Incisional Saline — Patient will be given a max of 30 cc injected through a 22g needle to area of incision.
  Arms: Saline
Drug: Post-Closure Local Anesthetic — Patient will be given a total of 0.5 mL/kg of 0.25% Bupivicaine either pre-incision: local will be to be given intradermally and onto the peritoneum under direct vision; or post-closure local will be injected intradermally after closure
  Other Names: Bupivicaine
  Arms: Local
Other: Post-Closure Saline — Patient will be given a max of 30 cc injected through a 22g needle after closing sutures were made.
  Arms: Saline

SUMMARY:
Patient will have usual appendectomy surgery with an injection of local or saline at incision site either before or after the incision at random.

The clinical hypothesis of this trial is that pediatric patients who undergo a local anesthetic pre-incisional and/or post-incisional will reduce the amount of postoperative pain and therefore reduce the amount of analgesics required to keep the patient satisfied.

Primary: To determine if local anesthetic reduces postoperative pain. Secondary: To assess the timing of local anesthetic injection affects postoperative pain.

DETAILED DESCRIPTION:
This is a prospective randomized-controlled pilot study of 100 pediatric subjects, recruited through Phoenix Children's Hospital and Pediatric Surgeons of Phoenix, who will undergo a laparoscopic appendectomy (LA) for acute non-perforated appendicitis. The reviewer and subject will be blind to the treatment to help prevent bias. The subjects will be randomized by envelope using a random number generator, and the infiltrated solution will be given to the surgeon by the pharmacy.

The subjects will be approached preoperatively and will be divided into three groups: pre-incisional injection of local anesthetic, post-incisional injection of local anesthetic, and (pre or post) injection of saline as the control.

All patients will have a standard 3 port laparoscopic appendectomy, port placement, port and instrument type, and operative technique will be determined by the surgeon's usual practice.

On induction, the following protocol will be utilized: a 2 mg/kg bolus of propofol, 1.5 mg/kg of lidocaine, 0.1 mg/kg of morphine, and 0.6 mg/kg of rocuronium. A standardized anesthetic, using a mixture of sevoflurane in oxygen and air, will be utilized. Once the appendectomy is complete, a single dose of 0.5 mg/kg of ketorolac will be given prior to extubation. A total of 0.5 mL/kg of 0.25% Bupivicaine or saline, up to a maximum of 30 cc, will be injected using a 22g needle. Pre-incision: local will be to be given intradermally and onto the peritoneum under direct vision; post-closure local will be injected intradermally after closure.

The subjects will be assessed for postoperative pain immediately upon wakening, and then 1, 2, 4, 8, 12, and 24 hours after the LA procedure by the bedside nurse by using the VAS and by measuring the total amount of opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Appendectomy for acute non-perforated appendicitis Must be between 9-17 years old

Exclusion Criteria:

* n/a

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Amount of Post Operative Pain Patients Experience | 12 hours
  The subjects will be assessed for post-operative pain immediately upon wakening, then at 1, 2, 4, 8, and 12 hours after procedure.

SECONDARY OUTCOMES:
The total amount of opioid use | 24 Hours
  This will be completed by looking at the total amount of morphine equivalants given to the patient during the first 24 hours of their hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addiss DG, Shaffer N, Fowler BS, Tauxe RV. The epidemiology of appendicitis and appendectomy in the United States. Am J Epidemiol. 1990 Nov;132(5):910-25. doi: 10.1093/oxfordjournals.aje.a115734. PMID 2239906
- [Background] Buckius MT, McGrath B, Monk J, Grim R, Bell T, Ahuja V. Changing epidemiology of acute appendicitis in the United States: study period 1993-2008. J Surg Res. 2012 Jun 15;175(2):185-90. doi: 10.1016/j.jss.2011.07.017. Epub 2011 Aug 9. PMID 22099604
- [Background] Edwards TJ, Carty SJ, Carr AS, Lambert AW. Local anaesthetic wound infiltration following paediatric appendicectomy: a randomised controlled trial: Time to stop using local anaesthetic wound infiltration following paediatric appendicectomy? Int J Surg. 2011;9(4):314-7. doi: 10.1016/j.ijsu.2010.09.012. Epub 2011 Feb 13. PMID 21324384
- [Background] Kang H, Kim BG. Intraperitoneal ropivacaine for effective pain relief after laparoscopic appendectomy: a prospective, randomized, double-blind, placebo-controlled study. J Int Med Res. 2010 May-Jun;38(3):821-32. doi: 10.1177/147323001003800309. PMID 20819419
- [Background] Liu Y, Seipel C, Lopez ME, Nuchtern JG, Brandt ML, Fallon SC, Manyang PA, Tjia IM, Baijal RG, Watcha MF. A retrospective study of multimodal analgesic treatment after laparoscopic appendectomy in children. Paediatr Anaesth. 2013 Dec;23(12):1187-92. doi: 10.1111/pan.12271. Epub 2013 Sep 25. PMID 24112856
- [Background] Masoomi H, Nguyen NT, Dolich MO, Mills S, Carmichael JC, Stamos MJ. Laparoscopic appendectomy trends and outcomes in the United States: data from the Nationwide Inpatient Sample (NIS), 2004-2011. Am Surg. 2014 Oct;80(10):1074-7. PMID 25264663
- [Background] Oravsky M, Bak V, Schnorrer M. Laparoscopic versus open appendectomy in treatment of acute appendicitis. Bratisl Lek Listy. 2014;115(10):660-2. doi: 10.4149/bll_2014_127. PMID 25573735
- [Background] Palmes D, Rottgermann S, Classen C, Haier J, Horstmann R. Randomized clinical trial of the influence of intraperitoneal local anaesthesia on pain after laparoscopic surgery. Br J Surg. 2007 Jul;94(7):824-32. doi: 10.1002/bjs.5810. PMID 17571296
- [Background] Reynolds SL, Jaffe DM. Diagnosing abdominal pain in a pediatric emergency department. Pediatr Emerg Care. 1992 Jun;8(3):126-8. doi: 10.1097/00006565-199206000-00003. PMID 1614900
- [Background] Scholer SJ, Pituch K, Orr DP, Dittus RS. Clinical outcomes of children with acute abdominal pain. Pediatrics. 1996 Oct;98(4 Pt 1):680-5. PMID 8885946
- [Background] Thanapal MR, Tata MD, Tan AJ, Subramaniam T, Tong JM, Palayan K, Rampal S, Gurunathan R. Pre-emptive intraperitoneal local anaesthesia: an effective method in immediate post-operative pain management and metabolic stress response in laparoscopic appendicectomy, a randomized, double-blinded, placebo-controlled study. ANZ J Surg. 2014 Jan-Feb;84(1-2):47-51. doi: 10.1111/j.1445-2197.2012.06210.x. Epub 2012 Oct 11. PMID 23057502
- [Background] Tomecka MJ, Bortsov AV, Miller NR, Solano N, Narron J, McNaull PP, Ricketts KJ, Lupa CM, McLean SA. Substantial postoperative pain is common among children undergoing laparoscopic appendectomy. Paediatr Anaesth. 2012 Feb;22(2):130-5. doi: 10.1111/j.1460-9592.2011.03711.x. Epub 2011 Sep 29. PMID 21958060
- [Background] Woolf CJ. Evidence for a central component of post-injury pain hypersensitivity. Nature. 1983 Dec 15-21;306(5944):686-8. doi: 10.1038/306686a0. PMID 6656869
- [Background] Wright JE. Controlled trial of wound infiltration with bupivacaine for postoperative pain relief after appendicectomy in children. Br J Surg. 1993 Jan;80(1):110-1. doi: 10.1002/bjs.1800800136. PMID 8428267